CLINICAL TRIAL: NCT05776329
Title: Randomized Controlled Clinical Trial on the Anti-inflammatory Effect of a Sustainable Dietary Strategy in Adults With Obesity
Brief Title: Dietary Intervention to Reduce Metabolic Endotoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Responsible Party: Principal Investigator, Silvia Yolanda Moya Camarena, Principal Investigator, Centro de Investigación en Alimentación y Desarrollo A.C.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SYMC001
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Endotoxemia; Intestinal Microbiota; Dietary Habits; Clinical Trial; Obesity
Keywords: Metabolic endotoxemia; Lipopolysaccharide binding protein; Dietary inflammatory index; Planetary health diet
MeSH Terms: conditions — Endotoxemia; Feeding Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: An interventional randomized controlled clinical trial of parallel design with active control.
Who Masked: Outcomes Assessor
Masking Description: Assignor to each group: The assignment of the people to the comparison groups will be carried out by the statistician responsible for the project. The statistician will not participate in any other project stage (registration, intervention, or measurements).
  Researcher in charge of the database: A person from outside the workgroup will assign codes to the participants enrolled in the study to prevent the person entering the data into the database from identifying the intervention group they belong to.
  Investigator in charge of the analysis of serum and stool samples: The same codes will be used to label the biological samples so that the person carrying out the interleukin and intestinal microbiota analyses cannot identify the intervention group to which they belong.
  The keys will be revealed at the end of the statistical analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-inflammatory and environmentally friendly dietary strategy (AIA-D) (Experimental): The environmentally friendly dietary strategy (AIA-D) designed based on the planetary health diet recommendations translated to the regional context and includes nutrients related to anti-inflammatory responses
  Interventions: Behavioral: AIA-D
- General healthy diet recommendations (CONV-D). (Active Comparator): The active comparator CONV-D is based on the general healthy diet recommendations
  Interventions: Behavioral: CONV-D

INTERVENTIONS:
Behavioral: AIA-D — The total energy contribution (1800 kcal/d) is 20% from protein, 25% from lipids, and 55% from carbohydrates. The recommendations include increasing protein intake primarily from plant sources, limiting the intake of red and processed meat, reducing refined sugar, and moderating dairy consumption. It also includes a list of locally produced and seasonal fruits and vegetables and a list of selected ingredients with anti-inflammatory properties to elaborate their foods. Participants will attend 3 motivational sessions of 1 h every two weeks. Besides nutrition and health, the motivational talks focused on the environmental impact of sustainability. Session 1: Planetary healthy diet. The inflammatory potential of diet. Explanation of the program. Session 2. Effect of ultra-processed food on health. Session 3. Healthy diets.
  Follow-up information, recipes, and pictures of dishes that meet the given recommendations will be sent once a week through closed social media groups.
  Arms: Low-inflammatory and environmentally friendly dietary strategy (AIA-D)
Behavioral: CONV-D — CONV-D is based on general healthy diet recommendations. The total energy contribution (1800 kcal/d) was 20% from protein, 25% from lipids, and 55% from carbohydrates.
  Among the recommended food groups are fruits (5 times a day), vegetables (5 times a day), cereals (3 times a day), legumes (3 times a day), dairy products (2 times a day), food of animal origin (3 times per day).
  Participants in the CONV-D group will attend one motivational and nutritional orientation session on day 1 of the intervention.
  Session 1. Food and nutrition. Obesity and diet. General healthy diet recommendations. Delivery of material (table of food equivalents).
  Follow-up information will be sent once a week through closed social media groups.
  Arms: General healthy diet recommendations (CONV-D).

SUMMARY:
The goal of this randomized clinical trial is to compare an antiinflammatory and environmentally friendly dietary strategy (AIA-D) designed based on the planetary health diet recommendations translated to the regional context and including nutrients related to antiinflammatory responses with an active control diet based on general healthy diet recommendations (CONV-D) in adults from 18 to 50 years of age with obesity (body mass index ≥30 kg/m2). The main questions it aims to answer are:

* If the intervention with AIA-D will cause a significant decrease at the end of the intervention (six weeks) in lipopolysaccharide-binding protein (LBP) compared to CONV-D.
* If intervention with AIA-D will cause a significant increase at the end of the intervention (six weeks) in the relative abundance of two specific bacteria genera (AM and FP) when compared to CONV-D.

Participants will:

* Sign the informed consent.
* Provide two peripheral blood samples (taken by our trained professionals).
* Provide two samples of feces.
* Allow anthropometric (body weight, height, hip and waist circumferences) blood pressure measurements on two occasions.
* Respond to 24 h dietary recall on two occasions.
* Attend the 1-hour group sessions requested (three for AIA-D and one for CONV-D).
* Follow the dietary recommendations provided.
* Be willing to participate in social media groups to receive information and follow up during the six weeks of the intervention.

Researchers will compare an antiinflammatory and environmentally friendly strategy (AIA-D) with an active control diet (CONV-D) based on general healthy diet recommendations to see if AIA-D decreases metabolic endotoxemia measured through LBP serum levels and increase the relative abundance of AM and FP, compared to CONV-D.

DETAILED DESCRIPTION:
This randomized clinical trial proposes to evaluate an environmentally friendly dietary strategy (AIA-D) designed based on the planetary health diet recommendations translated to the regional context and including nutrients related to anti-inflammatory responses that can decrease metabolic endotoxemia and promote FP and AM growth associated with anti-inflammatory effects and good intestinal health compared to an active control diet (CONV-D) general healthy diet recommendations.

Primary hypothesis: The intervention with a low-inflammatory and environmentally friendly dietary strategy aimed at adults diagnosed with obesity (body mass index ≥30 kg/m2) will cause a significant decrease at the end of the intervention (six weeks) in the levels of lipopolysaccharide-binding protein (metabolic endotoxemia), and significantly increase the relative abundance of AM and FP, when compared to general healthy diet recommendations.

Secondary hypotheses: The intervention with a low-inflammatory and environmentally friendly dietary strategy aimed at adults diagnosed with obesity (body mass index ≥30 kg/m2) will cause a significant increase at the end of the intervention (six weeks) in the relative abundance of Prevotella, when compared to general healthy diet recommendations.

The intervention with a low-inflammatory and environmentally friendly dietary strategy aimed at adults diagnosed with obesity (body mass index ≥30 kg/m2) will cause a significant decrease at the end of the intervention (six weeks) of body weight, percentage of body fat, body mass index, circumferences of waist and hip when compared to general healthy diet recommendations.

The intervention with a low-inflammatory and environmentally friendly dietary strategy aimed at adults diagnosed with obesity (body mass index ≥30 kg/m2) will improve blood pressure more than the general healthy diet recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Obesity according to body mass index: ≥ 30 kg/m2
* Willingness to participate and sign the consent form.
* Willingness to follow the dietary recommendations of the protocol.
* Have access to the internet and an electronic device.

Exclusion Criteria:

* Clinically diagnosed with hyperglycemia, hypertension, cardiovascular disease, renal disease, hepatic disease, immunosuppression, or another metabolic disease.
* Being under a dietary restriction regimen or pharmacological treatment to lose weight.
* Consuming dietary supplements for at least six months (vitamins, fatty acids, probiotics, prebiotics).
* Being under treatment with antibiotics or anti-inflammatory drugs in the last three months.
* Having bariatric surgery.
* Being pregnant or lactating.
* Present gastrointestinal disease
* Present Coronavirus disease (COVID-19) symptoms
* Develop diseases that affect body weight
* Becoming pregnant
* Withdrawal of informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Lipopolysaccharide-binding protein (LBP). | Baseline to six weeks
  Peripheral blood samples will be taken before and after the intervention, centrifuged for serum extraction, and stored at -80°C until analysis. ELISA kits were used to quantify LBP.
Change in relative abundance of FP | Baseline to six weeks
  According to the manufacturer's instructions, total DNA will be extracted from fecal samples and quantified by a spectrophotometer, where the ratio of 1.8-2.0 (260/280) is acceptable. DNA samples will be stored at -80°C until analysis. FP will be amplified from DNA extracted from fecal samples by quantitative polymerase chain reaction (qPCR). A specific set of primers will be used. The relative expression of the gen (relative abundance) will be calculated. The 16S ribosomal RNA (16S) (V4) normalizing gen will be used for analysis.
Change in relative abundance of AM | Baseline to six weeks
  According to the manufacturer's instructions, total DNA will be extracted from fecal samples and quantified by a spectrophotometer, where the ratio of 1.8-2.0 (260/280) is acceptable. DNA samples will be stored at -80°C until analysis. AM will be amplified from DNA extracted from fecal samples by quantitative polymerase chain reaction (qPCR). A specific set of primers will be used. The relative expression of the gen (relative abundance) will be calculated. The 16S ribosomal RNA (16S) (V4) normalizing gen will be used for analysis.

SECONDARY OUTCOMES:
Change in abundance of Prevotella | Baseline to six weeks
  According to the manufacturer's instructions, total DNA will be extracted from fecal samples and quantified by a spectrophotometer, where the ratio of 1.8-2.0 (260/280) is acceptable. DNA samples will be stored at -80°C until analysis. Prevotella will be amplified from DNA extracted from fecal samples by quantitative polymerase chain reaction (qPCR). A specific set of primers will be used. The relative expression of the gen (relative abundance) will be calculated. The 16S ribosomal RNA (16S) (V4) normalizing gen will be used for analysis.
Change in body weight | Baseline to six weeks
  Body weight will be measured with minimal clothing using a digital electronic scale (capacity of 0 to 150 ± 0.05 kg).
Change in body mass index | Baseline to six weeks
  The body mass index will be calculated by dividing the weight (kg) by the square of height (m). Height will be measured using a stadiometer (rank 0.70-2.05 m) while barefoot participants were standing with their heads in the Frankfurt plane
Change in hip circumference | Baseline to six weeks
  The hip circumference will be measured using a flexible anthropometric tape (200 cm) at the widest circumference of the gluteus.
Change in waist circumference | Baseline to six weeks
  The waist circumference will be measured using a flexible anthropometric tape (200 cm) at the level of the umbilicus
Change in waist-to-hip ratio | Baseline to six weeks
  The waist-to-hip ratio will be calculated by dividing waist circumference (cm) by hip circumference (cm).
Change in percentage of body fat | Baseline to six weeks
  An electrical bioimpedance analysis device will measure body fat.
Change in the dietary inflammatory index. | Baseline to six weeks
  The DII and energy-adjusted-DII (E-DII) will be calculated from the dietary data collected using 24-h dietary recall for each participant. E-DII scores were calculated using the density approach wherein all nutrients were converted to 1000 kcal consumption.
Change in blood pressure | Baseline to six weeks
  Systolic and diastolic blood pressure will be measured by a digital device.
Retention | Baseline to six weeks
  Percentage of participants that finished the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Y Moya-Camarena, Ph. D., Principal Investigator — Centro de Investigación en Alimentación y Desarrollo
Locations (2):
- Mexico (2):
  - Universidad Vizcaya de las Américas, Hermosillo, Sonora
  - Centro de Investigación en Alimentación y Desarrollo, Hermosillo, Sonora

IPD SHARING:
Plan to Share IPD: No
The database will be available from the principal investigator upon reasonable request.

REFERENCES:
- [Background] Halmos EP, Christophersen CT, Bird AR, Shepherd SJ, Gibson PR, Muir JG. Diets that differ in their FODMAP content alter the colonic luminal microenvironment. Gut. 2015 Jan;64(1):93-100. doi: 10.1136/gutjnl-2014-307264. Epub 2014 Jul 12. PMID 25016597
- [Background] Gray L, Hasebe K, O'Hely M, Ponsonby AL, Vuillermin P, Collier F; BIS Investigator Group. Rapid PCR identification of Prevotella copri in an Australian cohort of pregnant women. J Dev Orig Health Dis. 2020 Jun;11(3):228-234. doi: 10.1017/S2040174419000849. Epub 2019 Dec 17. PMID 31843036
- [Background] Shivappa N, Steck SE, Hurley TG, Hussey JR, Hebert JR. Designing and developing a literature-derived, population-based dietary inflammatory index. Public Health Nutr. 2014 Aug;17(8):1689-96. doi: 10.1017/S1368980013002115. Epub 2013 Aug 14. PMID 23941862
- [Background] Hebert JR, Shivappa N, Wirth MD, Hussey JR, Hurley TG. Perspective: The Dietary Inflammatory Index (DII)-Lessons Learned, Improvements Made, and Future Directions. Adv Nutr. 2019 Mar 1;10(2):185-195. doi: 10.1093/advances/nmy071. PMID 30615051
- [Background] Willett W, Rockstrom J, Loken B, Springmann M, Lang T, Vermeulen S, Garnett T, Tilman D, DeClerck F, Wood A, Jonell M, Clark M, Gordon LJ, Fanzo J, Hawkes C, Zurayk R, Rivera JA, De Vries W, Majele Sibanda L, Afshin A, Chaudhary A, Herrero M, Agustina R, Branca F, Lartey A, Fan S, Crona B, Fox E, Bignet V, Troell M, Lindahl T, Singh S, Cornell SE, Srinath Reddy K, Narain S, Nishtar S, Murray CJL. Food in the Anthropocene: the EAT-Lancet Commission on healthy diets from sustainable food systems. Lancet. 2019 Feb 2;393(10170):447-492. doi: 10.1016/S0140-6736(18)31788-4. Epub 2019 Jan 16. No abstract available. PMID 30660336